CLINICAL TRIAL: NCT02547363
Title: Efficacy and Safety of LEO 43204 in Field Treatment of Actinic Keratosis on Balding Scalp Including 12-month Follow-up
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP0084-1195
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Results first posted 2018-12-26 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2018-12

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEO 43204 (Experimental): Treatment once daily for 3 days
  Interventions: Drug: LEO 43204 gel
- Vehicle gel (Placebo Comparator): Treatment once daily for 3 days
  Interventions: Drug: Vehicle gel

INTERVENTIONS:
Drug: LEO 43204 gel
  Other Names: Ingenol Disoxate
  Arms: LEO 43204
Drug: Vehicle gel
  Arms: Vehicle gel

SUMMARY:
The objective of the trial is to compare the short term efficacy of LEO 43204 gel with vehicle gel in AK on the balding scalp when applied topically once daily for 3 consecutive days as field treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with 5 to 20 clinically typical, visible and discrete AKs within a treatment area of sun-damaged skin on the full balding scalp (the balding part of the scalp should be greater than 25 cm2 (4 in2) and up to approximately 250 cm2 (40 In2)
* Subjects with minimum 3 clinically typical, visible and discrete AKs within a tracking area of 50 cm2 (8 In2). The tracking area must be within the treatment area

Exclusion Criteria:

* Location of the treatment area (full balding scalp) within 5 cm of an incompletely healed wound or within 5 cm of a suspected BCC or SCC
* Treatment with ingenol mebutate gel in the treatment area within the last 12 months
* Lesions in the treatment area that have: atypical clinical appearance (e.g. hyperthrophic, hyperkeratotic or cutaneous horns) and /or, recalcitrant disease (e.g. did not respond to cryotherapy on two previous occasions)
* History or evidence of skin conditions other than the trial indication that would interfere with the evaluation of the trial medication (e.g. eczema, unstable psoriasis, xeroderma pigmentosum)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2015-11; Primary Completion 2016-08-17 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Siegel, MD, Principal Investigator — Long Island Skin Center
Locations (1):
- Long Island Skin Cancer & Dermatologic Surgery, Smithtown, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 373 participants were enrolled, 57 were screening failures, and 316 participants were randomized. Only 313 of the randomized participants were treated with investigational medicinal product (IMP), the number of participants treated is reflected as the number of participants started in the first period.
Groups:
- LEO 43204 0.037% Gel: Treatment once daily with LEO 43204 0.037% gel for 3 consecutive days applied on the scalp.
- Vehicle Gel: Treatment once daily with vehicle gel for 3 consecutive days applied on the scalp.
Period: 3-day Treatment and 8-week Follow-up
Arm/Group | LEO 43204 0.037% Gel | Vehicle Gel
Started | 211 | 105
Treated | 209 | 104
Completed | 207 | 94
Not Completed | 4 | 11
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 2 | 8
Not completed — Lost to Follow-up | 1 | 1
Not completed — Other | 1 | 1
Period: 12-month Follow-up
Arm/Group | LEO 43204 0.037% Gel | Vehicle Gel
Started | 204 | 86
Completed | 194 | 81
Not Completed | 10 | 5
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 4 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- LEO 43204 0.037% Gel: Treatment once daily for 3 days with LEO 43204 0.037% gel
- Vehicle Gel: Treatment once daily for 3 days with vehicle gel
- Total: Total of all reporting groups
Arm/Group | LEO 43204 0.037% Gel | Vehicle Gel | Total
Number analyzed (Participants) | 209 | 104 | 313
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (9.1) | 69.9 (9.3) | 70.5 (9.2)
Age, Customized [Count of Participants; unit: Participants]
  Age group: 18-64 years | 45 | 28 | 73
  Age group: 65-84 years | 155 | 70 | 225
  Age group: >=85 years | 9 | 6 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 208 | 104 | 312
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 69 | 37 | 106
  France | 13 | 7 | 20
  United Kingdom | 18 | 9 | 27
  United States | 109 | 51 | 160

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Clearance of Actinic Keratosis (AK)
Description: The number of clinically visible actinic keratosis lesions (AKs) identified in the treatment area was recorded at Day 1 (baseline), Week 4 and Week 8.
  Complete clearance was defined as no clinically visible AKs in the treatment area.
Time Frame: At Week 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LEO 43204 0.037% Gel | Vehicle Gel
Number analyzed (Participants) | 209 | 104
percentage of participants | 25.8 [20.4 to 32.2] | 0.0 [0.0 to 3.6]
Statistical Analysis 1: Comparison: LEO 43204 0.037% Gel vs Vehicle Gel; Test type: Superiority; p < 0.001, Fisher exact test

2. Secondary Outcome: Percentage of Participants With Partial Clearance of AKs
Description: Partial clearance was defined as at least 75% reduction from baseline in the number of clinically visible AKs in the treatment area.
Time Frame: At Week 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LEO 43204 0.037% Gel | Vehicle Gel
Number analyzed (Participants) | 209 | 104
percentage of participants | 58.9 [52.1 to 65.3] | 1.0 [0.2 to 5.2]
Statistical Analysis 1: Comparison: LEO 43204 0.037% Gel vs Vehicle Gel; The p-values for secondary endpoints have been corrected by the Holm-Bonferroni method to account for multiplicity. The prespecified multiplicity adjustment by the Holm-Bonferroni method requires the ordering of the p-values for the secondary endpoints by size; Test type: Superiority; p < 0.001, Mantel Haenszel; Ratio of clearance rates = 62.59, 95% CI 2-sided [8.68 to 451.08] — Mantel-Haenszel estimate (0.037% relative to vehicle), adjusted for pooled sites

3. Secondary Outcome: Percentage of Participants With Partial Clearance of AKs
Description: as for outcome 2
Time Frame: At Week 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LEO 43204 0.037% Gel | Vehicle Gel
Number analyzed (Participants) | 209 | 104
percentage of participants | 57.4 [50.6 to 63.9] | 1.0 [0.2 to 5.2]
Statistical Analysis 1: Comparison: LEO 43204 0.037% Gel vs Vehicle Gel; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Mantel Haenszel; Ratio of clearance rates = 59.21, 95% CI 2-sided [8.44 to 415.35] — Mantel-Haenszel estimate (0.037% relative to vehicle), adjusted for pooled sites

4. Secondary Outcome: Percent Reduction in AK Count in the Treatment Area Compared to Baseline
Description: The percent reduction at Week 8 from baseline was analysed using a negative binomial regression for the AK count at Week 8 with treatment group and pooled sites as factors and baseline count as offset variable. The table presents adjusted mean percent reduction at Week 8 from baseline.
Time Frame: At Week 8
Measure: Mean (95% Confidence Interval); unit: percentage of reduction
Arm/Group | LEO 43204 0.037% Gel | Vehicle Gel
Number analyzed (Participants) | 209 | 104
percentage of reduction | 72.3 [69.1 to 75.2] | -2.0 [-16.0 to 10.3]
Statistical Analysis 1: Comparison: LEO 43204 0.037% Gel vs Vehicle Gel; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Mantel Haenszel; Week 8 AK count ratio = 0.27, 95% CI 2-sided [0.23 to 0.32] — 0.037% relative to vehicle

ADVERSE EVENTS:
Time Frame: Treatment period including follow-up (from Day 1 to Week 8) and extended follow-up (from Week 8 up to Month 14)
Description: Adverse events presented in the table are investigator-reported terms. Adverse events of special interest within system organ class (SOC) Neoplasm benign, malignant and unspecified (incl cysts and polyps), were adjudicated by an Independent Adjudication Committee based on central biopsy review.
  For further details on the adjudication outcomes, see link to the full report in section "More information" Adverse events are reported with a >=2% frequency threshold for the active treatment group.
Groups:
- LEO 43204 0.037% Gel - Extended Follow-up: Treatment once daily for 3 days with LEO 43204 0.037% gel
- Vehicle Gel - Extended Follow-up: Treatment once daily for 3 days with vehicle gel
Arm/Group | LEO 43204 0.037% Gel | Vehicle Gel | LEO 43204 0.037% Gel - Extended Follow-up | Vehicle Gel - Extended Follow-up
Serious Adverse Events (participants affected / at risk) | 4/209 | 2/104 | 1/204 | 0/86
Other Adverse Events (participants affected / at risk) | 153/209 | 9/104 | 18/204 | 12/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LEO 43204 0.037% Gel (N=209) | Vehicle Gel (N=104) | LEO 43204 0.037% Gel - Extended Follow-up (N=204) | Vehicle Gel - Extended Follow-up (N=86)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0 | 0
Neoplasm of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LEO 43204 0.037% Gel (N=209) | Vehicle Gel (N=104) | LEO 43204 0.037% Gel - Extended Follow-up (N=204) | Vehicle Gel - Extended Follow-up (N=86)
Periorbital oedema (Eye disorders) | 14 | 0 | 0 | 0
Application site discomfort (General disorders) | 6 | 2 | 0 | 0
Application site injury (General disorders) | 8 | 0 | 0 | 0
Application site pain (General disorders) | 127 | 3 | 0 | 0
Application site pruritus (General disorders) | 64 | 2 | 0 | 0
Application site scar (General disorders) | 1 | 1 | 10 | 7
Face oedema (General disorders) | 5 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 6 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 5 | 1
Headache (Nervous system disorders) | 21 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 5 | 0 | 0 | 0
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO acknowledges the investigators right to publish the entire results of the study, irrespective of outcome. LEO retains the right to have any publication submitted to LEO for review. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.